CLINICAL TRIAL: NCT05112679
Title: Limb Health and Socket Pressure in Response to Powered Ankle Prostheses
Brief Title: Limb Health and Socket Pressure in Response to Powered Ankle Protheses
Acronym: OPORP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Notre Dame (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Sashwati Roy, Professor of Surgery, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 12350
Record Dates: First submitted 2021-08-13; First posted 2021-11-09 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pressure Ulcer, Ankle; Prosthesis User; Prosthesis Durability; Mobility Limitation; Skin Wound; Amputation; Traumatic, Foot; Amputation; Limb Deficiencies
MeSH Terms: conditions — Pressure Ulcer; Prosthesis Failure; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Proprio Foot (Experimental): each participant was randomized to use Proprio or empower based on randomization followed by switching the other empower or proprio
  Interventions: Device: PROPRIO FOOT® by Ossur & Empower ankle by Ottobock
- Empower foot (Experimental): ach participant was randomized to use Proprio or empower based on randomization followed by switching the other empower or proprio
  Interventions: Device: PROPRIO FOOT® by Ossur & Empower ankle by Ottobock

INTERVENTIONS:
Device: PROPRIO FOOT® by Ossur & Empower ankle by Ottobock — PROPRIO FOOT is a microprocessor controlled foot that offer great potential to more completely restore the locomotor capabilities of individuals with transtibial amputation, Empower: Empower powered ankle offer great potential to more completely restore the locomotor capabilities of individuals with transtibial amputation.

SUMMARY:
this project seeks to understand and quantify the effects of powered transtibial prostheses on socket loading and direct measures of residual limb health so as to inform the optimization of prosthesis fit.

DETAILED DESCRIPTION:
Some estimates suggest that by 2050, as many as 3.6 million people in the United States will be living with limb loss, and at least 60% of them will have had at least a foot removed For military personnel, combat-related amputations remain one of the most common major disabling war-related injuries from modern armed conflict. Technological advancements in active prosthetic devices for individuals with transtibial amputation offer the potential for superior function in key areas that could lead to higher rates of RTD and improved quality of life. Currently intended primarily for individuals with a K-level of 3 or 4, active transtibial prostheses that provide controlled plantar/dorsiflexion in either swing (microprocessor-controlled prostheses) or late stance (prostheses with powered propulsion) are likely to become the gold standard in the future as technology continues to improve Indeed, users of these types of prostheses have higher mobility than those using any of the other four categories of prosthetic ankle-foot mechanisms for unlimited community ambulators. Note that a major insurer has recently declared microprocessor-controlled ankle-foot prostheses medically necessary for members whose functional level is 3 or above.The PROPRIO FOOT® by Ossur, is a microprocessor-controlled prosthesis that regulates the angle of ankle dorsiflexion during the swing phase. This added ankle control of these devices reduces the risk of falls by increasing toe clearance supports more natural standing posture on slopes and improves stair and slope ascent/descent capability by adapting to the change in terrain. On stairs, the PROPRIO FOOT® has been shown to improve affected leg knee kinematics (increased knee flexion) and kinetics (increased knee moment) instance. These improvements also contributed to higher interlimb symmetry reduced energetic cost of slope ascent and higher Amputee Mobility Predictor with a Prosthesis (AMPPRO) scores . Although the ankle of the PROPRIO FOOT® can be controlled in swing, the device does not have adequate power to provide an active propulsion instance. The Empower ankle by Ottobock is a powered prosthesis that provides active propulsion in late stance to mimic the positive work performed by the ankle plantar flexors in push-off. The Empower has been shown to improve affected leg kinematics (increased ankle range of motion and reduced knee flexion) on smooth flat ground ramp ascent and gravel]. In terms of kinetics, the Empower likewise results in increased ankle power on level ground stairs and ramps . Active prostheses like the PROPRIO FOOT® and Empower ankle offer great potential to more completely restore the locomotor capabilities of individuals with transtibial amputation, perhaps enhancing RTD for military personnel. As with all prosthetic components, though, these active devices are of little use if they induce pain and/or injury at the residual limb to the degree that the user will simply not wear them. The investigators will examine how optimal fit of lower limb prostheses can impact individuals comfort and/or reduce irritation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and above
* Weight ≤ 280 lb
* Ambulate at a K3 level or higher-level determined from patient EHR
* At least 3 months post-amputation per physician discretion
* Residual limb length greater than 4.5 inches
* Use of a passive prosthesis
* Unilateral transtibial amputees
* Must be able to ambulate without any assistive devices
* Subjects must be able to follow directions and give informed consent on their own

Exclusion Criteria:

* Conditions and/or co-morbidities that would prevent wearing a prosthetic socket, affect gait, or influence function of the contralateral limb
* Other amputees
* Cognitive deficits or mental health problems that would limit ability to consent and participate fully in the study protocol
* Women who are pregnant or who plan to become pregnant in the near future
* Individuals diagnosed with renal failure
* Participants unwilling to wear a cloth face covering for the duration of each visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share deidentified patient data consisting of the patient PEQ and comfort scores and transpepidermal water loss data upon request.
Supporting Information: SAP, ICF
Time Frame: 6 months after completion
Access Criteria: Email study contact

RESULTS

PARTICIPANT FLOW:
Groups:
- Proprio Foot, Then Empower Ankle: Participants started with the PROPRIO FOOT® by Ossur, a microprocessor-controlled prosthesis that regulates the angle of ankle dorsiflexion during the swing phase. After four weeks of use, participants crossed over to use the Empower ankle by Ottobock, an active powered ankle prosthesis, for an additional four weeks.
- Empower Ankle, Then Proprio Foot: Participants started with the Empower ankle by Ottobock, an active powered ankle prosthesis. After four weeks of use, participants crossed over to use the PROPRIO FOOT® by Ossur, a microprocessor-controlled prosthesis that regulates the angle of ankle dorsiflexion during the swing phase, for an additional four weeks.
Period: Overall Study
Arm/Group | Proprio Foot, Then Empower Ankle | Empower Ankle, Then Proprio Foot
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: all participants that have completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Proprio Foot, Then Empower Ankle | Empower Ankle, Then Proprio Foot | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6
participants completed the study visits [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Powered Transtibial Prosthesis on Socket Pressure
Description: effects of a powered transtibial prosthesis on the socket pressure for level-ground walking to a microprocessor-controlled prosthesis and a passive prosthesis
Time Frame: 4 weeks
Population: accurate in-socket pressure data could be only collected from 3 subjects
Measure: Mean (Standard Deviation); unit: kPa/kg
Groups:
- Proprio Foot: Participants who used the PROPRIO FOOT® by Ossur, a microprocessor-controlled prosthesis that regulates the angle of ankle dorsiflexion during the swing phase, for four weeks.
- Empower Ankle: Participants who used the Empower ankle by Ottobock, an active powered ankle prosthesis, for four weeks.
Arm/Group | Proprio Foot | Empower Ankle
Number analyzed (Participants) | 3 | 3
kPa/kg | 0.58 (0.01) | 0.25 (0.03)
Statistical Analysis 1: Comparison: Proprio Foot vs Empower Ankle; All participants were randomized to both groups in a cross over design, if a participant started with proprio after 4 weeks of use they will cross over to Empower ankle or vice versa. the data reflect comparison of the groups; Test type: Other — See SAP; p = 0.009, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.007, Standard Deviation 0.21

2. Secondary Outcome: Change in Skin Perfusion
Description: Changes measured with laser speckle imaging. The perfusion data is expressed as perfusion units (PU) which is a dimensionless ratio calculated by dividing the standard deviation of the intensity in a given area by the mean intensity within that area, essentially representing the degree of variation in the speckle pattern. Higher number indicates greater perfusion which is better outcome.
Time Frame: 4 weeks
Population: accurate data only from n=4 participants were obtained in Empower foot.
Measure: Mean (Standard Deviation); unit: Perfusion Units (PU)
Arm/Group | Proprio Foot | Empower Ankle
Number analyzed (Participants) | 6 | 4
Perfusion Units (PU) | 1.1 (0.75) | 0.8 (0.7)

3. Secondary Outcome: Transepidermal Water Loss (TEWL)
Description: Water loss change is measured via the TEWL device- the lower score mean a better outcome for TEWL.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: g/m^2 x h
Arm/Group | Proprio Foot | Empower Ankle
Number analyzed (Participants) | 6 | 5
g/m^2 x h | 2.0 (0.61) | 0.8 (0.21)

ADVERSE EVENTS:
Time Frame: period of all study visits from baseline (week 0) to final visit (week 8); each intervention was evaluated for four weeks
Arm/Group | Proprio Foot | Empower Ankle
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT05112679/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT05112679/ICF_000.pdf